CLINICAL TRIAL: NCT06823414
Title: Endoscopy/Robotic Assisted Nipple Skin Sparing Mastectomy and Inmediate Reconstruction With Prepectoral Implant. Prospective Study for the Evaluation of the Feasibility and Safety of the Technique, Quality of Life and Cosmetic Results
Brief Title: Endoscopy/Robotic Assisted Nipple Skin Sparing Mastectomy
Status: Recruiting | Type: Observational
Sponsor: Alejandra García-Novoa (Other)
Responsible Party: Sponsor-Investigator, Alejandra García-Novoa, Principal Investigator, University Hospital A Coruña
Organization: University Hospital A Coruña (Other)
Other Study IDs: VideoBreast-24
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Cancer Non-invasive Breast Cancer; High Risk Breast Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Video assisted mastectomy: Patients with a video-assisted nipple skin sparing mastectomy
  Interventions: Other: Video assisted mastectomy

INTERVENTIONS:
Other: Video assisted mastectomy — Nipple Skin sparing mastectomy assisted by endoscopic or robotic

SUMMARY:
Non-inferiority study of video-assisted (endoscopic or robotic) skin- and nipple-sparing mastectomy compared to open mastectomy. The feasibility of the technique, oncological safety and cosmetic results will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Women who require a mastectomy and who do not require skin reduction or resection are included. Women with both breast cancer and those at high risk for breast cancer are included.

Exclusion Criteria:

* Sarcomas of the breast.
* Benign breast tumors.
* Prepectoral reconstruction with expansion.
* Impossibility to preserve the skin.
* Need for reduction pattern
* Inability to perform an MRI during follow-up (obesity, claustrophobia, etc.).
* Inability to complete the BREAST-Q™ questionnaire due to the patient's cognitive alterations.
* Refusal of the patient to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patient with breast cancer or high risk for breast cancer who need a mastectomy. The mastectomy will be skin and nipple preserving and will be performed with endoscopic assistance
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
Implant Loss | First year after surgery
  Safety of the reconstruction technique, calculated by the number of implants lost

SECONDARY OUTCOMES:
local relapse | first 5 years
  evaluate oncological safety in terms of local relapses
Glandular residual tissue | first year
  Residual glandular tissue after endoscopic mastectomy identified by magnetic resonance imaging one year after the intervention
Suvival | 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Unit. First floor. Hospital Abente y Lago. Paseo del General Sir John Moore, 4, A Coruña, Galicia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] 1. Acea-Nebril B, García-Novoa A, Cereijo-Garea C, Conde C, Bouzón A, Díaz C. Safety and Quality of Life in Women with Immediate Reconstruction with Polyurethane Implants after Neoadjuvant Chemotherapy: Outcomes from The Preq-20 Trial. Cancers 2023;15(4):1113. doi: 10.3390/cancers15041113. 2. Acea B, García A, García L, Díaz C, Bouzón A, Conde C. Immediate breast reconstruction by prepectoral polyurethane implant: Preliminary results of the prospective study PreQ-20. Cir Esp (Engl Ed) 2023;101(3):187-197. doi: 10.1016/j.cireng.2022.09.021. 3. Nakajima H, Sakaguchi K, Mizuta N, et al. Video-assisted total glandectomy and immediate reconstruction for breast cancer. Biomed Pharmacother 2002;56 Suppl 1:205s-8s. 4. Wei Ch, Lai HW. Endoscopic-assisted surgery in the management of breast cancer: 20 years review of trend, techniques and outcomes. Breast; 2019:46:144-156. doi: 10.1016/j.breast.2019.05.013. 5. Wei Ch, Lai HW. Evolution of minimal access breast surgery. Gland Surg 2019;8(6):784-793. doi: 10.21037/gs.2019.11.16. 6. Toesca A, Paradze N, Manconi A, Galimberti V, Intra M, Colleoni M et al. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast 2017; Feb:31:51-56. doi: 10.1016/j.breast.2016.10.009. 7. Rathat G, Herlin C, Bonnel C, Captier G, Duraes M. Endoscopic Nipple-Sparing Mastectomy with Immediate Prepectoral Implant-Based Reconstruction: A Case Report Am J Case Rep 2019;20:1812-1816. doi: 10.12659/AJCR.919669.